CLINICAL TRIAL: NCT00288444
Title: Defining the Interaction of Docetaxel and Lonafarnib in Patients With Advanced Malignancies
Brief Title: Interaction of Docetaxel and Lonafarnib in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Aventis Pharmaceuticals (Industry); Schering-Plough (Industry)
Responsible Party: Principal Investigator, John Kauh, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 174-2004; EU841-03
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Lung Cancer; Soft Tissue Sarcoma; Colorectal Carcinoma; Breast Cancer; Prostate Cancer
Keywords: Advanced malignancies.
MeSH Terms: conditions — Lung Neoplasms; Sarcoma; Colorectal Neoplasms; Breast Neoplasms; Prostatic Neoplasms | interventions — lonafarnib; Docetaxel

ARMS (4):
- Docetaxel 36 mg/ m2 IV weekly and Lonafarnib 150 mg (Active Comparator): Docetaxel 36 mg/ m^2 Intravenously weekly and Lonafarnib 150 mg by mouth twice a day daily.
  Interventions: Drug: Lonafarnib; Drug: Docetaxel
- Docetaxel 30 mg/ m2and Lonafarnib 150 mg (Active Comparator): Docetaxel 30 mg/ m^2 Intravenously weekly and Lonafarnib 150 mg by mouth twice a day daily.
  Interventions: Drug: Lonafarnib; Drug: Docetaxel
- Docetaxel 36 mg/ m2 and Lonafarnib 100 mg (Active Comparator): Docetaxel 36 mg/ m^2 Intravenously weekly and Lonafarnib 100 mg by mouth twice a day daily
  Interventions: Drug: Lonafarnib; Drug: Docetaxel
- Docetaxel 30 mg/m2 and Lonafarnib 100 mg (Active Comparator): Docetaxel30 mg/m^2 Intravenously weekly and Lonafarnib 100 mg by mouth twice a day daily.
  Interventions: Drug: Lonafarnib; Drug: Docetaxel

INTERVENTIONS:
Drug: Lonafarnib
  Other Names: SCH66336
Drug: Docetaxel
  Other Names: Taxotere

SUMMARY:
To determine the molecular interaction in tumor samples between docetaxel and lonafarnib.

DETAILED DESCRIPTION:
1. To determine the safety and toxicity of intravenous docetaxel, administered on a weekly schedule (3 weeks out of 4), in combination with oral lonafarnib, administered on a daily schedule, in patients with locally advanced and metastatic solid tumor malignancies which are refractory to the standard of care.
2. To determine the pharmacokinetic interaction between docetaxel and lonafarnib.
3. To determine the molecular interaction in peripheral blood mononuclear cells between docetaxel and lonafarnib

ELIGIBILITY:
Inclusion Criteria:.1.1 Patient must have a pathologically-confirmed locally advanced or metastatic solid tumor malignancy demonstrated to be refractory to the standard of care, with tumors accessible by needle or surgical biopsy.

3.1.2 Only patients determined to be at minimal risk to receiving the biopsy (with tumor location/accessibility as well as underlying patient comorbidities judged to allow a minimal risk biopsy by the radiologist/surgeon performing the procedure) will be eligible for this study.

3.1.3 Patient must have an ECOG performance status of 2 or less.

3.1.4 Patient must have a life-expectancy of at least 12 weeks.

3.1.5 Patient must have adequate bone marrow function: WBC ≥ 3,000 cells/mm3, ANC ≥ 1,500 cells/mm3, platelet count ≥ 100,000/mm3 and Hgb ≥ 9.0 g/dL.

3.1.6 Patient must have adequate liver function: total bilirubin level ≤ 2.0 mg/dL and ≤ ULN, albumin ≥ 2.5 g/dL.

3.1.7 Patient must have adequate renal function: Transaminases/Alkaline phosphatase: AST or ALT and alkaline phosphatase must be within the range allowing for eligibility. This range is defined as ≤ 2 x ULN.

In determining eligibility, the more abnormal of the two (AST or ALT) should be used.

3.1.8 Patient must have received no more than three previous chemotherapy regimens (prior chemotherapy may or may not have contained a taxane).

3.1.9 Patient must meet the specified informed consent requirement.

3.1.10 Patient must be of age ≥ 18 years.

3.1.11 Women of childbearing age must have a negative pregnancy test.

3.1.12 Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

3.1.13 Patient must have ≤ Grade 1 neurotoxicity from previous anticancer treatment or from any cause.

3.1.14 Patient must have adequate coagulation function: INR and PTT ≤ 1.5 x ULN.

3.1.15 Patient must have discontinued all prior chemotherapy and radiotherapy at least 4 weeks prior to registration.

3.1.16 Patient must have discontinued use of the following drugs which are an inducers or inhibitors of CYP3A4 at least 2 days prior to registration: ethinylestradiol, gestodene, itraconazole, ketoconazole, cimetidine, erythromycin, carbamazepine, high dose chronic steroids, phenobarbital, phenytoin, rifampin (rifampcin), and sulfinpyrazone.

Patient must have a pathologically-confirmed

-

Exclusion Criteria:

3.2.1 Patient has received more than three previous chemotherapy regimens.

3.2.2 Patient is pregnant or breast feeding.

3.2.3 Patient has signs of symptoms of acute infection requiring systemic therapy.

3.2.4 Patient exhibits confusion, disorientation, or has a history of major psychiatric illness which may impair the patient's understanding of the informed consent.

3.2.5 Patient's life expectancy is less than 12 weeks.

3.2.6 Patient has > Grade 1 neurotoxicity from previous anticancer treatment or significant neuropathy from any cause.

3.2.7 Patient requires total parenteral nutrition with lipids.

3.2.8 Inability to swallow the lonafarnib BID.

3.2.9 Patient has a history of uncontrolled heart disease (including clinically significant coronary artery disease, congestive heart failure and symptomatic or uncontrolled arrythmias).

3.2.10 Patient has a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80. Symptoms include: any reaction such as bronchospasm, generalized urticaria, systolic BP ≤ 80mm Hg, and angioedema.

3.2.11 Use of chronic steroids or anticonvulsants.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Determine the molecular interaction | Four weeks

SECONDARY OUTCOMES:
Determine safety and efficacy | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Kauh, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Winship Cancer Institute, Atlanta, Georgia, United States